CLINICAL TRIAL: NCT04921592
Title: Neuromodulation Training for Upper Extremity Recovery for Chronic Cervical Spinal Cord Injury
Brief Title: Upper Extremity Training for Chronic Cervical Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Gail Forrest, Director, Center for Spinal Stimulation, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R-1153-21
Record Dates: First submitted 2021-05-12; First posted 2021-06-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized into 1 of 3 groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transcutaneous stimulation (Experimental): 1. transcutaneous stimulation 60 sessions
  2. Transcutaneous stimulation 40sessions
  3. Transcutaneous stimulation 20 sessions
  Interventions: Other: upper extremity stimulation

INTERVENTIONS:
Other: upper extremity stimulation — transcutaneous stimulation of the upper extremities
  Other Names: Activity-Based Recovery Therapy (ABRT)

SUMMARY:
This study is to understand how the combination of activity-based recovery training and targeted spinal cord transcutaneous stimulation (scTS) can improve participants' ability to use their hand, arms, and core.

DETAILED DESCRIPTION:
This study is to understand how the combination of activity-based recovery training and targeted spinal cord transcutaneous stimulation (scTS) can improve participants' ability to use their hand, arms, and core. Activity-based recovery training aims to advance independence without the use of assistive devices. Spinal cord transcutaneous stimulation is an electrical stimulation that is provided on top of the skin over specific areas of the spinal cord to activate the circuitry for the activity that is being trained and reconnect with pathways between the brain and spinal cord.

i) Physical evaluation by the clinician or physician including the Classification of Spinal Cord Injury (ISNCSCI exam. ii) A series of tests to evaluate the trunk, arm function with and without using tests to evaluate muscle activation. iii) A series of questionnaires to evaluate function and quality of life iv) Two separate Magnetic Resonance Imaging (MRI) of spinal column (head to hip).

Randomized to one of three groups:

Group 1: will be upper extremity training with transcutaneous spinal stimulation of the spine combined with upper extremity and trunk rehabilitation. The group will complete 60 training sessions transcutaneous spinal stimulation.

Group 2: will be upper extremity training with transcutaneous spinal stimulation of the spine combined with upper extremity and trunk rehabilitation. The group will complete 40 training sessions of transcutaneous spinal stimulation. The group will then complete 20 sessions of rehabilitation therapy of the upper extremities and trunk (no stimulation).

Group 3: will be will be upper extremity training with transcutaneous spinal stimulation of the spine combined with upper extremity and trunk rehabilitation. The group will complete 20 training sessions of transcutaneous spinal stimulation. The group will then complete 40 sessions of rehabilitation therapy of the upper extremities and trunk (no stimulation).

Transcutaneous spinal stimulation will involve stimulating the spinal segments between C5/6 to lumber regions. Training time will be approximately 1 hour, 3-4 times per week.

Rehabilitation therapy will involve exercises concentrating on fingers, hand, arm and trunk function. A physical therapist will be at training and testing sessions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age.
* spinal cord injury for greater than or equal to 6 months.
* spinal cord injury at a cervical neurologic level of injury.

Exclusion Criteria:

* ventilator dependent.
* history of fractures.
* pressure sore or skin issues.
* history of illicit drug abuse.
* history of cardiac, respiratory, bladder, renal or other medical disorder unrelated to spinal cord injury.
* bladder Botox injections less than 12 months prior.
* muscle Botox injections less than 12 months prior.
* colostomy bag or urostomy.
* implanted pump (i.e., baclofen pump, pain pump, etc).
* If I am female: I am pregnant at the time of enrollment or planning to become pregnant during the course of the study.
* unable to wean from anti-spasticity medication.
* contraindications to MRI imaging (pacemaker, metallic foreign body, aneurysm clip, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Neuro Recovery Scale ( NRS). | 6 months
  Measure of the degree a person who has sustained a spinal cord injury (SCI) has recovered the ability to perform functional tasks relative to how the individual performed these tasks prior to injury. The NRS consists of a numeric version of the visual analog scale. The most common form of the NRS is a horizontal line with an eleven point numeric range. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible. This type of scale can be administered verbally.

CONTACTS AND LOCATIONS:
Overall Officials: Gail F Forrest, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No